CLINICAL TRIAL: NCT03911921
Title: Renshen Yangrong Tang (RSYRT) for Reducing Fatigue in Cancer Survivors: A Phase II Randomized Trial
Brief Title: RSYR for Fatigue Reduction in Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yichen Xu, Research leader, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FATIGUE; PZ2017019 (Other Grant/Funding Number: Beijing Municipal Hospital Administration Training Program)
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cancer-related Problem/Condition
Keywords: Fatigue, Cancer
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Huang Qi

STUDY DESIGN:
Intervention Model Description: a randomized Phase II trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSYYT decoction (Experimental): RSYYT decoction Compound granules of traditional Chinese medicine
  Interventions: Drug: RSYRT decoction
- Astragalus membranaceus (Experimental): one herb decoction Compound granules of one herb (Astragalus membranaceus)
  Interventions: Drug: Astragalus membranaceus

INTERVENTIONS:
Drug: RSYRT decoction — Compound granules of traditional Chinese medicine
  Arms: RSYYT decoction
Drug: Astragalus membranaceus — One herb
  Arms: Astragalus membranaceus

SUMMARY:
This randomized Phase II trial to establish the efficacy of traditional Chinese medicine (TCM) herbal products above control group for treating fatigue in patients with cancer.

DETAILED DESCRIPTION:
Patients who were randomized and been enrolled in, had stable disease and no anemia, and reported moderate to severe fatigue over two months (rated ≥4 on a 0-10 scale). Patients took TCM decoction Renshen Yangrong decoction (RSYR),Which containing 12 TCM herbs, twice a day for 6 weeks. RSYRT aims to correct Qi deficiency. Fatigue was assessed before and after RSYRT therapy.

ELIGIBILITY:
Inclusion Criteria:

Pathological diagnosis of malignant tumors; 3 months without surgery, radiotherapy and chemotherapy, biological treatment; Hemoglobin > 11g/L; Complete remission of the lesion, or recent review of the Disease is stable, the estimated survival time is more than 6 months; ECOG score is 0-2, fatigue score of the last 24 hours > 4 ; Age is 18-65 years old; TCM syndrome differentiation for deficiency of qi; Liver, kidney function, electrolyte normal; Willing to join the group and sign the informed consent.

Exclusion Criteria:

Allergies to herbs and plant drugs; Uncontrollable diabetes, hypertension, TSH abnormalities, uncontrollable pain, and a history of myocardial infarction within 6 months; Scores of anxiety disorders and depression (HAD-D) were 11 or more, antidepressants and antioxidants were used in the past month; Breast cancer receptor positive patients took endocrine therapy drugs; Tonics were used in the past 2 weeks.; Children, pregnant and lactating women; Receiving anemia-related treatment; Chinese medicine syndrome differentiation with excessive heat; Unable to read or understand the scale.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Fatigue score | 6 weeks
  Self-assessed 24-hour fatigue symptom score. According to the NCCN fatigue guide, the score is 0-10 points, 0 points means no fatigue, 10 points means the most serious fatigue that can be imagined.

CONTACTS AND LOCATIONS:
Overall Officials: Pingping Li, Prof., Study Director — Peking University Cancer Hospital & Institute; Ting Lu, Dr., Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu Y, Wang XS, Chen Y, Shi Q, Chen TH, Li P. A Phase II Randomized Controlled Trial of Renshen Yangrong Tang Herbal Extract Granules for Fatigue Reduction in Cancer Survivors. J Pain Symptom Manage. 2020 May;59(5):966-973. doi: 10.1016/j.jpainsymman.2019.10.018. Epub 2019 Oct 24. PMID 31668965